CLINICAL TRIAL: NCT05899049
Title: An Open-label, Randomized Phase 3 Study to Evaluate Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Belzutifan (MK-6482) and Lenvatinib (MK-7902), or MK-1308A in Combination With Lenvatinib, Versus Pembrolizumab and Lenvatinib, as First-Line Treatment in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Study of Pembrolizumab (MK-3475) in Combination With Belzutifan (MK-6482) and Lenvatinib (MK-7902), or Pembrolizumab/Quavonlimab (MK-1308A) in Combination With Lenvatinib, vs Pembrolizumab and Lenvatinib, for Treatment of Advanced Clear Cell Renal Cell Carcinoma (MK-6482-012)-China Extension Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-012 China Extension; MK-6482-012 China Extension (Other: MSD); jRCT2031210435 (Registry Identifier: jRCT(Japan Registry of Clinical Trials)); PHRR210911-003887 (Registry Identifier: Philippine Health Research Registry (PHRR))
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Hypoxia inducible factor (HIF); Hypoxia inducible factor 1B (HIF-1B); Hypoxia inducible factor 2 alpha (HIF-2 alpha)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; belzutifan; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Pembrolizumab + Belzutifan + Lenvatinib (Experimental): Participants will receive pembrolizumab 400 mg PLUS belzutifan 120 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered intravenously (IV) once every 6 weeks (Q6W) for up to 18 administrations (up to ~2 years). Belzutifan and lenvatinib will be administered orally once daily (QD) until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Belzutifan; Drug: Lenvatinib
- Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants will receive pembrolizumab/quavonlimab (co-formulation of pembrolizumab 400 mg and quavonlimab 25 mg) PLUS lenvatinib 20 mg. Pembrolizumab/quavonlimab will be administered IV Q6W for up to 18 administrations (up to ~2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab/Quavonlimab; Drug: Lenvatinib
- Pembrolizumab + Lenvatinib (Active Comparator): Participants will receive pembrolizumab 400 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered IV Q6W for up to 18 administrations (up to ~2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 400 mg administered Q6W via IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Belzutifan + Lenvatinib; Pembrolizumab + Lenvatinib
Drug: Belzutifan — Belzutifan 120 mg administered QD via oral tablet
  Other Names: MK-6482; PT2977; WELIREG™
  Arms: Pembrolizumab + Belzutifan + Lenvatinib
Biological: Pembrolizumab/Quavonlimab — Pembrolizumab/quavonlimab is a co-formulated product composed of pembrolizumab 400 mg in combination with quavonlimab 25 mg, administered Q6W via IV infusion
  Other Names: MK-1308A
  Arms: Pembrolizumab/Quavonlimab + Lenvatinib
Drug: Lenvatinib — Lenvatinib 20 mg administered QD via oral capsule
  Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
The goal of this China extension study is to evaluate the efficacy and safety of pembrolizumab plus belzutifan plus lenvatinib or pembrolizumab/quavonlimab plus lenvatinib versus pembrolizumab plus lenvatinib as first-line treatment in Chinese participants with advanced clear cell renal cell carcinoma (ccRCC).

The primary hypotheses are (1) pembrolizumab plus belzutifan plus lenvatinib is superior to pembrolizumab plus lenvatinib with respect to progression-free survival (PFS) and overall survival (OS), in advanced ccRCC participants; and (2) pembrolizumab/quavonlimab plus lenvatinib is superior to pembrolizumab plus lenvatinib with respect to PFS and OS, in advanced ccRCC participants.

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-6482-012 (NCT04736706) plus those enrolled during the China extension enrollment period. A total of approximately 249 Chinese participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of RCC with clear cell component.
* Has received no prior systemic therapy for advanced ccRCC
* Male participants are abstinent from heterosexual intercourse or agree to use contraception during and for at least 7 days after last dose of study intervention with belzutifan and lenvatinib.
* Female participants are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) or use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after pembrolizumab or pembrolizumab/quavonlimab or for at least 30 days after last dose of lenvatinib or belzutifan, whichever occurs last
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function.
* Participants receiving bone resorptive therapy must have therapy initiated at least 2 weeks prior to randomization/allocation

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has had major surgery, other than nephrectomy within 4 weeks prior to randomization
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has received prior radiotherapy within 2 weeks prior to first dose of study intervention
* Has hypoxia or requires intermittent supplemental oxygen or requires chronic supplemental oxygen
* Has clinically significant cardiac disease within 12 months from first dose of study intervention
* Has a history of interstitial lung disease
* Has symptomatic pleural effusion; a participant who is clinically stable following treatment of this condition is eligible
* Has preexisting gastrointestinal or non-gastrointestinal fistula
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has a known psychiatric or substance abuse disorder that would interfere with requirements of the study
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study drug; killed vaccines are allowed
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of noninfectious pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B
* Has radiographic evidence of intratumoral cavitation, encasement or invasion of a major blood vessel
* Has clinically significant history of bleeding within 3 months prior to randomization
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 58 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR based on RECIST 1.1 will be presented.
Overall Survival (OS) | Up to approximately 58 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 58 months
  ORR is defined as the percentage of participants who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by BICR based on RECIST 1.1 will be presented.
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 58 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by BICR based on RECIST 1.1 will be presented.
Number of Participants Who Experienced At least One Adverse Event (AE) | Up to approximately 58 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 58 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- China (17):
  - Beijing Cancer hospital-Renal carcinoma and melanoma ( Site 6000), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 6009), Chongqing, Chongqing Municipality
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 6003), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University-Urology ( Site 6036), Guangzhou, Guangdong
  - Guangzhou First People's Hospital ( Site 6007), Guangzhou, Guangdong
  - Henan Cancer Hospital-Urology ( Site 6006), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 6002), Wuhan, Hubei
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( S, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University-Urology ( Site 6025), Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 6019), Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 6014), Xi'an, Shaanxi
  - West China Hospital Sichuan University-Urology Surgery ( Site 6016), Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University ( Site 6032), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 6024), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing ( Site 6033), Jiaxing, Zhejiang
  - Ningbo First Hospital-Urology ( Site 6028), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Urology Surgery ( Site 6021), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/